CLINICAL TRIAL: NCT07255053
Title: Comparative Effects of Post Isometric Relaxation and Post Facilitation Stretching on Pain Reduction Hip Abduction and Internal Rotation Range, and Functional Disability in Patients With Piriformis Syndrome
Brief Title: Comparative Effects of PIR and PFS on Pain, Hip ROM, and Disability in Piriformis Syndrome
Acronym: PIR-PFS RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Aqsa Bashir, Dr, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUF-PIRIFORMIS-RCT-2025
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups: Post-Isometric Relaxation or Post-Facilitation Stretching, and interventions are delivered in parallel
Masking Description: Open-label study; participants, care providers, and investigators are aware of the assigned interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post Isometric Relaxation (PIR) (Experimental): Type of technique: Muscle Energy Technique (MET)
  Patient position: Supine, affected leg flexed at hip and knee, crossed over the other leg, foot resting on the table
  Pelvis stabilization: Therapist hand on opposite ASIS to prevent pelvic movement
  Leg positioning: Other hand on lateral aspect of the knee
  Finding the barrier: Knee moved into abduction until first sign of resistance (pain-free end range)
  Isometric contraction: Patient pushes against the therapist's hand at ~20% strength for 7-10 seconds
  Relaxation and stretch: After contraction, leg moved slightly further into abduction
  Repetitions: 3 times per session
  Interventions: Procedure: Post Isometric Relaxation (PIR)
- Post Facilitation Stretching (PFS) (Experimental): Patient position: Supine, affected leg slightly adducted and externally rotated, hip flexed >60°
  Therapist hand placement: Inferior hand on table for support, superior hand guides leg movement
  Muscle positioning: Piriformis placed in intermediate range (between full stretch and rest)
  Isometric contraction: Patient externally rotates leg against resistance for 10 seconds
  Pause / Rest phase: 30-second relaxation after contraction; therapist applies deeper stretch into adduction and external rotation
  Next barrier: Leg gently moved to new barrier
  Repetitions: 3 times per session
  Interventions: Procedure: Post Facilitation Stretching (PFS)

INTERVENTIONS:
Procedure: Post Isometric Relaxation (PIR) — Participants received PIR exercises targeting the piriformis muscle three days per week for 4 weeks. The technique involved pain-free isometric contractions followed by gentle stretching to improve hip abduction and internal rotation
  Other Names: Muscle Energy Technique (MET)
  Arms: Post Isometric Relaxation (PIR)
Procedure: Post Facilitation Stretching (PFS) — Participants received PFS exercises targeting the piriformis muscle three days per week for 4 weeks. The technique combined isometric contractions with controlled stretching to enhance hip mobility and reduce pain.
  Other Names: Muscle Energy Technique (MET)
  Arms: Post Facilitation Stretching (PFS)

SUMMARY:
This randomized clinical trial evaluates the effectiveness of Post-Isometric Relaxation (PIR) and Post-Facilitation Stretching (PFS) for managing pain, improving hip abduction and internal rotation, and enhancing functional capacity in patients with Piriformis Syndrome. Thirty-six participants will be assessed at baseline and six weeks using pain scores, hip range of motion, and functional scales to determine which technique provides superior outcomes.

DETAILED DESCRIPTION:
Piriformis Syndrome (PS) is a musculoskeletal condition characterized by pain in the buttock and hip, sometimes radiating to the lower back and thigh. It may arise from anatomical variations affecting the sciatic nerve, inflammation, hypertrophy, muscle spasms, or shortening of the piriformis muscle. PS can significantly reduce hip range of motion and functional capacity, affecting patients' quality of life.

This randomized clinical trial aimed to compare the effectiveness of two rehabilitation techniques, Post-Isometric Relaxation (PIR) and Post-Facilitation Stretching (PFS), in managing pain, improving hip abduction and internal rotation, and enhancing functional capacity in patients with PS. Thirty-six participants aged 35-55 years, of both genders, diagnosed with sub-acute or chronic PS, and meeting specific clinical criteria, were randomly assigned to either intervention group.

Inclusion criteria included positive findings on at least three of the following tests: Piriformis, Beatty, Freiberg, FAIR, Sign of Pace, and Nagel tonic external rotation of hip; bilateral buttock pain due to sciatic nerve or piriformis muscle spasm; NPRS pain score of 3-7; tenderness over the sciatic foramen; and willingness to participate. Exclusion criteria included spinal, hip, knee, or SI joint pathology, prior spinal surgery or vertebral fracture, systemic disease, limb length discrepancy, postural deformities (e.g., scoliosis), hip dislocation or femoral fracture, and any psychological conditions.

Group A (PIR) participants performed exercises lying supine with the affected leg flexed, pelvis stabilized, and piriformis muscle activated through resisted abduction. Group B (PFS) participants performed combined stretching and isometric contractions with the involved leg positioned in hip flexion, adduction, and external rotation. Interventions were conducted over a 4-week period.

Assessments were conducted at baseline and six weeks using:

Numeric Pain Rating Scale (NPRS) to quantify pain intensity

Goniometer - to measure hip abduction and internal rotation range

Lower Extremity Functional Scale (LEFS) to assess functional disability; a 20-item scale rated on a Likert scale (total score 0-80), with lower scores indicating greater disability

The objective of this study was to determine which rehabilitation technique, PIR or PFS, is more effective in alleviating pain, improving hip range of motion, and enhancing functional outcomes, ultimately aiming to improve the quality of life for patients diagnosed with Piriformis Syndrome.

ELIGIBILITY:
Inclusion Criteria:

- Participants aged 35-55 years Both genders Positive findings on three or more of the following tests: Piriformis, Beatty, Freiberg, FAIR, Sign of Pace, Nagel tonic external rotation of hip Bilateral buttock pain caused by compression of the sciatic nerve or piriformis muscle spasm NPRS pain score between 3 and 7 Tenderness to palpation over the sciatic foramen Diagnosed sub-acute or chronic Piriformis Syndrome Willing to participate

Exclusion Criteria:

* Any pathology or recent injury around the hip, knee, or SI joint, or radiating pain from the spine, SI joint, or hip History of spinal surgery or vertebral fracture History of systemic disease, stroke, leprosy, or amputation Leg pain not related to Piriformis Syndrome (e.g., disc herniation, sacroiliac joint dysfunction, degenerative joint disease) History of spinal injury, joint disease, or congenital abnormalities Limb length difference SI joint dysfunction Hip joint dislocation or femoral fracture Any postural deformity or anomaly (e.g., scoliosis) Psychologically diagnosed condition

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Pain intensity in patients with Piriformis Syndrome | Baseline and 4 weeks after intervention completion
  Pain was measured using the Numeric Pain Rating Scale (NPRS), a 0-10 scale where 0 indicates no pain and 10 indicates worst possible pain.

SECONDARY OUTCOMES:
Hip Abduction and Internal Rotation Range of Motion | Baseline and 4 weeks after intervention completion
  Hip range of motion was measured using a goniometer to assess internal rotation and abduction angles.
Functional Disability | Baseline and at 4 weeks after intervention completion
  Functional capacity was assessed using the Lower Extremity Functional Scale (LEFS), a 20-item questionnaire evaluating lower limb function in daily activities. Lower scores indicate greater disability

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Faisalabad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data from this study, including pain scores (NPRS), hip range of motion (internal rotation and abduction), and functional scores (LEFS), will be shared with qualified researchers upon reasonable request. The shared data will be used for secondary analyses, meta-analyses, and reproducibility studies related to Piriformis Syndrome interventions.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available 6 months after publication of the main results and will remain available for 5 years after study completion
Access Criteria: Data will be shared with researchers who submit a methodologically sound proposal and agree to use data only for the stated purpose. Access will require signing a Data Use Agreement (DUA)